CLINICAL TRIAL: NCT00625404
Title: Phase 3, Multi-center, Double-blind, Randomized, Placebo-controlled Effectiveness and Safety Study to Assess the Role of Truvada® in Preventing HIV Acquisition in Women
Brief Title: FEM-PrEP (Truvada®): Study to Assess the Role of Truvada® in Preventing HIV Acquisition in Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10015
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: HIV Infections
Keywords: Aspartate Aminotransferase (AST); Alanine Aminotransferase (ALT); HIV; HIV Prevention; Oral PrEP; Truvada; women; Tenofovir; TDF; FTC; emtricitabine; hepatitis; Pre-exposure Prophylaxis (PrEP); HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Hepatitis | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Truvada Arm (Experimental): Daily single oral tablet of Truvada (TDF/FTC), a fixed-dose combination of emtricitabine (FTC; 200 mg) and tenofovir disoproxil fumarate (TDF; 300 mg).
  Interventions: Drug: Truvada
- Placebo Arm (Placebo Comparator): Daily single oral tablet of Placebo. Tablets are identical to Truvada tablets in taste and appearance; however, they contain no active ingredients.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Truvada — Daily single oral tablet of Truvada - a fixed-dose combination of emtricitabine (FTC; 200 mg) and tenofovir disoproxil fumarate (TDF; 300 mg).
  Other Names: TDF/FTC - emtricitabine and tenofovir disoproxil fumarate
  Arms: Truvada Arm
Other: Placebo — Daily single oral tablet of Placebo. Tablets are identical to Truvada tablets in taste and appearance; however, they contain no active ingredients.
  Arms: Placebo Arm

SUMMARY:
This Phase III, double-blind, randomized, placebo-controlled trial enrolled HIV-negative women from 4 sites in 3 countries (Kenya, Tanzania, South Africa). The study's purpose was to investigate the safety and effectiveness of a once-daily Truvada® pill (compared with placebo) in preventing HIV among HIV-uninfected women at risk of becoming infected through sexual intercourse.

The study population included HIV-antibody-negative women between the ages of 18-35 who were at risk of HIV acquisition through sexual intercourse. Each participant was randomized to take either a daily single oral tablet of Truvada®, which is a fixed-dose combination of emtricitabine (FTC; 200 mg) and tenofovir disoproxil fumarate (TDF; 300 mg), or an identical placebo.

After enrollment, each participant was followed every four weeks. All participants were followed for an additional eight weeks after study drug was stopped. Incidence rates of HIV infection were compared between the two groups (active drug and placebo) using the intent-to-treat principle.

DETAILED DESCRIPTION:
This Phase III, double-blind, randomized, placebo-controlled trial enrolled HIV-negative women from 4 sites in 3 countries (Kenya, Tanzania, South Africa). The study's purpose was to investigate the safety and effectiveness of a once-daily Truvada® pill (compared with placebo) in preventing HIV among HIV-uninfected women at risk of becoming infected through sexual intercourse.

The study population included HIV-antibody-negative women between the ages of 18-35 who were at risk of HIV acquisition through sexual intercourse. Each participant was randomized to take either a daily single oral tablet of Truvada®, which is a fixed-dose combination of emtricitabine (FTC; 200 mg) and tenofovir disoproxil fumarate (TDF; 300 mg), or an identical placebo. All participants received risk reduction counseling and condoms. Women had to be using a study-approved effective non-barrier contraceptive method at the time of enrollment and were asked to do so for the whole period they were on study drug. They received contraceptive counseling throughout the study. Any diagnosed, treatable sexually transmitted infection was treated free of charge.

After enrollment, each participant was followed every four weeks. All participants were followed for an additional eight weeks after study drug was stopped. Participants at risk for Hepatitis B Virus (HBV) flare were followed every four weeks for 12 weeks after stopping study product. Participants who acquired HIV infection during the study stopped taking the study drug at the time of HIV diagnosis, and will be followed for 52 weeks post diagnosis and were referred for care and treatment. Participants who became pregnant stopped taking the study drug but continued follow-up visits. Incidence rates of HIV infection were compared between the two groups (active drug and placebo) using the intent-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able (see criterion 2) to provide written informed consent to be screened for and to participate in the trial
2. Able to answer a percentage of informed consent screening (75%) and enrollment (100%) comprehension quiz questions correctly
3. Between 18-35 years old, inclusive
4. At higher risk of becoming HIV infected
5. Have a final negative result according to the site-specific screening HIV testing algorithm and a final negative result at enrollment according to the study HIV testing algorithm
6. Willing to participate in all aspects of the study and to comply with study procedures, for up to 60 weeks, including:

   * Be randomized
   * Use study product as directed
   * Adhere to follow-up schedule and willing to be contacted by site staff between study visits (by phone and/or in person)
   * Use a study-approved effective non-barrier method of contraception for the duration of the study
   * Take study product, as evidenced by swallowing a vitamin tablet that is similar in size to the study product at enrollment
   * Provide contact information and agrees to some form of contact method throughout the study
7. Not intending to relocate out of the area for the duration of the study participation and does not have a job or other obligations that may require long absences from the area ( > 1 month at a time)
8. In general good health and have no condition (social or medical) which, in the opinion of the Site Investigator, would make study participation unsafe or complicate data interpretation
9. Not pregnant or breastfeeding, and does not anticipate a desire for pregnancy during the 52 weeks of on-product participation
10. Medically eligible at screening including:

    * Adequate renal function (serum creatinine ≤ upper limit of normal (ULN) of local range and creatinine clearance ≥ 60ml/min estimated by the Cockcroft-Gault Creatinine Clearance Formula
    * Adequate hepatic function (hepatic transaminases ALT and AST < 2x ULN [according to local normal ranges])
    * HBsAg negative
    * Serum phosphorus levels above the lower limit of the local normal range (according to local normal ranges - grade 3 & 4 hypophosphatemia will be excluded even if within normal local ranges)
11. Not received or receiving an experimental HIV vaccine, participating in another HIV prevention study or participating in any other clinical trial with a biomedical intervention
12. No clinical signs of liver disease (e.g., ascites, spider angiomata, hepatomegaly, jaundice)
13. No definite evidence of glycosuria or proteinuria (i.e., no repeated positive [ ≥ + 1 ] urine dipstick). If a urine dipstick is positive for either glucose and/or protein at the first test, a second urine sample will be tested.
14. No history of pathological bone fractures
15. No history of adverse reaction to latex
16. Not taking any of the following medications: nephrotoxic agents; aminoglycoside antibiotics (including gentamicin); intravenous (IV) amphotericin B; cidofovir; cisplatin; foscarnet; IV pentamidine; oral or IV vancomycin; oral or IV gancyclovir; other agents with significant nephrotoxic potential; drugs that slow renal excretion; probenecid; immune system modulators; systemic chemotherapeutic agents (i.e. cancer treatment medications); systemic corticosteroids; interleukin-2 (IL-2); immunomodulators; interferon (alpha, beta, or gamma); other antiretrovirals (including nucleoside analogs, non-nucleoside reverse transcriptase inhibitors, protease inhibitors or investigational antiretroviral agents)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2120 (Actual)
Dates: Start 2009-05; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lut Van Damme, MD, MS, PhD, Principal Investigator — FHI 360; Amy Corneli, PhD, MPH, Principal Investigator — FHI 360; Jennifer Deese, MPH, Study Director — FHI 360
Locations (4):
- Bondo Clinic, Bondo District Hospital, Bondo, Nyanza, Kenya
- South Africa (2):
  - Setshaba Research Centre, Pretoria, Gauteng
  - Josha Research Center, Bloemfontein
- Arusha Clinic, Levolosi Health Center, Arusha, Tanzania

REFERENCES:
- [Result] Lut Van Damme, M.D., Amy Corneli, Ph.D. and Douglas Taylor, Ph.D. New England Journal of Medicine 367: 411-422, 2012
- [Derived] Mandala J, Nanda K, Wang M, De Baetselier I, Deese J, Lombaard J, Owino F, Malahleha M, Manongi R, Taylor D, Van Damme L. Liver and renal safety of tenofovir disoproxil fumarate in combination with emtricitabine among African women in a pre-exposure prophylaxis trial. BMC Pharmacol Toxicol. 2014 Dec 24;15:77. doi: 10.1186/2050-6511-15-77. PMID 25539648
- [Derived] Grant RM, Liegler T, Defechereux P, Kashuba AD, Taylor D, Abdel-Mohsen M, Deese J, Fransen K, De Baetselier I, Crucitti T, Bentley G, Agingu W, Ahmed K, Damme LV. Drug resistance and plasma viral RNA level after ineffective use of oral pre-exposure prophylaxis in women. AIDS. 2015 Jan 28;29(3):331-7. doi: 10.1097/QAD.0000000000000556. PMID 25503265
- [Derived] Todd CS, Deese J, Wang M, Hubacher D, Steiner MJ, Otunga S, Van Damme L; FEM-PrEP Study Group. Sino-implant (II)(R) continuation and effect of concomitant tenofovir disoproxil fumarate-emtricitabine use on plasma levonorgestrel concentrations among women in Bondo, Kenya. Contraception. 2015 Mar;91(3):248-52. doi: 10.1016/j.contraception.2014.10.008. Epub 2014 Oct 22. PMID 25459097
- [Derived] Van Damme L, Corneli A, Ahmed K, Agot K, Lombaard J, Kapiga S, Malahleha M, Owino F, Manongi R, Onyango J, Temu L, Monedi MC, Mak'Oketch P, Makanda M, Reblin I, Makatu SE, Saylor L, Kiernan H, Kirkendale S, Wong C, Grant R, Kashuba A, Nanda K, Mandala J, Fransen K, Deese J, Crucitti T, Mastro TD, Taylor D; FEM-PrEP Study Group. Preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2012 Aug 2;367(5):411-22. doi: 10.1056/NEJMoa1202614. Epub 2012 Jul 11. PMID 22784040
- See also: Genetics Home Reference for complement factor I deficiency — http://ghr.nlm.nih.gov/condition/complement-factor-i-deficiency
- See also: MedlinePlus: AIDS — http://www.nlm.nih.gov/medlineplus/hivaids.html
- See also: MedlinePlus: Hepatitis — http://www.nlm.nih.gov/medlineplus/hepatitis.html
- See also: Drug Information: n-Octadecanoic acid — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0000057114&QV1=N-OCTADECANOIC+ACID
- See also: Drug Information: Calcium stearate — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0001592230&QV1=CALCIUM+STEARATE
- See also: Drug Information : Aluminum monostearate — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0007047849&QV1=ALUMINUM+MONOSTEARATE
- See also: U.S. FDA Resources — http://clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Groups:
- Truvada Arm: Daily single oral tablet of Truvada, a fixed-dose combination of emtricitabine (FTC; 200 mg) and tenofovir disoproxil fumarate (TDF; 300 mg).
Period: Overall Study
Arm/Group | Truvada Arm | Placebo Arm
Started | 1062 | 1058
Completed | 855 | 885
Not Completed | 207 | 173

BASELINE CHARACTERISTICS:
Groups:
- Truvada Arm; Placebo Arm: Daily single oral tablet of Placebo. Tablets are identical to Truvada tablets in taste and appearance; however, they contain no active ingredients.
- Total: Total of all reporting groups
Arm/Group | Truvada Arm | Placebo Arm | Total
Number analyzed (Participants) | 1062 | 1058 | 2120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1062 | 1058 | 2120
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 23 (18-35) [18 to 35] | 23 (18-35) [18 to 35] | 23 (18-35) [18 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1062 | 1058 | 2120
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: HIV Infection
Description: HIV Seroconversion, with time to infection refined based on PCR results obtained from stored specimens.
Time Frame: Cumulative HIV infection between enrollment and 52 weeks
Population: All randomized participants who made at least one follow-up visit and were not HIV-positive at enrollment were included in the analysis population
Measure: Number; unit: participants
Groups:
- Truvada Arm; Placebo Arm: The effectiveness population consisted of all women who were randomized and who had at least one follow-up visit and were not HIV PCR positive at enrollment. This population consisted of 2056 women (1024 in the Truvada arm, 1032 in the placebo arm) and was used for baseline analyses.
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 1024 | 1032
participants | 33 [3.25 to 6.63] | 35 [3.47 to 6.93]
Statistical Analysis 1: Comparison: Truvada Arm vs Placebo Arm; Hazard ratio (HR) for HIV infection based on proportional hazards model, stratified on site. Study was designed to have 90% power to reject the null hypothesis that the HR for infection is > 0.3; Test type: Superiority or Other; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.59 to 1.52]

2. Primary Outcome: Confirmed Grade 2 or Higher Serum Creatinine Toxicity
Description: Repeat specimens were collected to confirm chemistry toxicities. Grade 2 or higher serum creatinine toxicity was defined as ≥1.4 times the upper limit of normal
Time Frame: cumulative toxicity through 52 weeks of product use and 4 weeks post product
Population: The Safety Population consisted of all women who were randomized and who had at least one follow-up visit and did not return all of their product un-used. Only women assessed for a particular safety outcome were included in analysis of that outcome.
Measure: Number; unit: participants
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 1021 | 1033
participants | 4 | 2
Statistical Analysis 1: Comparison: Truvada Arm vs Placebo Arm; Log-rank test for difference in rate of grade 2 or higher creatinine, based on time to first event; Test type: Superiority or Other; p = 0.45, Log Rank

3. Primary Outcome: Frequency of Adverse Events (AEs) During and Within 4 Weeks After Study Product Administration
Description: The total number of adverse events in the placebo and Truvada arms during and within 4 weeks after study product administration.
Time Frame: 10-26 months per site
Population: The Safety Population, a subset of the ITT Population, excludes participants who never received study product, returned all product unused, or never returned for a follow-up visit. Analyses were performed by randomly assigned treatment group.
Measure: Number; unit: Number of adverse events
Groups:
- Truvada Arm; Placebo Arm: The Safety Population, a subset of the ITT Population, excludes participants who never received study product, returned all product unused, or never returned for a follow-up visit. Analyses were performed by randomly assigned treatment group.
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 1025 | 1033
Number of adverse events | 2257 | 2384

4. Primary Outcome: Confirmed Grade 3 or Higher Reduction in Phosphorus
Description: Repeat specimens were collected to confirm chemistry toxicities. Grade 3 phosphorus reduction was defined as ≤2.4mg/dL
Time Frame: Through 52 weeks on product and 4 weeks post-product
Measure: Number; unit: participants
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 1021 | 1033
participants | 45 | 40
Statistical Analysis 1: Comparison: Truvada Arm vs Placebo Arm; Log-rank test for difference in rates between groups; Test type: Superiority or Other; p = 0.59, Log Rank

5. Primary Outcome: Confirmed Grade 3 or Higher ALT Elevation
Description: Grade 3 or higher ALT elevation was defined as ≥ 2.6 times the upper limit of normal
Time Frame: Through 52 weeks on product and 4 weeks post-product
Measure: Number; unit: participants
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 1021 | 1033
participants | 6 | 8
Statistical Analysis 1: Comparison: Truvada Arm vs Placebo Arm; Log-rank test for difference in rates between groups; Test type: Superiority or Other; p = 0.79, Log Rank

6. Primary Outcome: Confirmed Grade 3 or Higher AST Elevation
Description: Grade 3 or higher AST elevation was defined as ≥ 2.6 times the upper limit of normal
Time Frame: Through 52 weeks on product and 4 weeks post-product
Measure: Number; unit: participants
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 1021 | 1033
participants | 3 | 1
Statistical Analysis 1: Comparison: Truvada Arm vs Placebo Arm; Log-rank test for difference in rates between groups; Test type: Superiority or Other; p = 0.62, Log Rank

7. Secondary Outcome: Plasma HIV RNA Level (HIV-1 Viral Load)
Description: Viral load at the time of HIV detection, HIV conversion and through 16 weeks
Time Frame: up to 16 weeks
Population: 68 women who became infected post-enrollment were included in viral load analyses. Only 48 of these women (27 on Truvada and 21 on placebo) contributed a specimen sample for analysis at the 16-weeks post seroconversion visit
Measure: Log Mean (Standard Deviation); unit: log copies/mL
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 27 | 21
log copies/mL | 4.40 (1.05) | 4.37 (1.08)
Statistical Analysis 1: Comparison: Truvada Arm vs Placebo Arm; t-test for difference on viral loads; Test type: Superiority or Other; p = 0.89, t-test, 2 sided; Mean Difference (Final Values) = 0.03

8. Secondary Outcome: CD4+ T-cell Count
Description: CD4+ T-cell Count at the Time of HIV Seroconversion through 16 weeks
Time Frame: Up to 16 weeks
Measure: Mean (Standard Deviation); unit: cells/mL
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 26 | 20
cells/mL | 579.3 (318.2) | 601.4 (318.5)
Statistical Analysis 1: Comparison: Truvada Arm vs Placebo Arm; t-test for difference in mean CD-4 counts; Test type: Superiority or Other; p = 0.82, t-test, 2 sided; Mean Difference (Final Values) = 22.1

9. Secondary Outcome: FTC and/or Tenofovir Resistance
Description: Genotypic resistance to FTC and/or tenofovir at the time of HIV diagnosis and 4 weeks later. If resistance was present, testing was repeated at weeks 12, 24, 36 and 52 as necessary (resistance testing will stop if no resistance is detected).
  participants were classified as having resistance if they had one or more visits in which resistance was detected, even if the resistance became undetectable over time.
Time Frame: up to 52 weeks
Population: All women who seroconverted were assessed for possible resistance.
Measure: Number; unit: participants
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 33 | 35
participants | 3 | 1

10. Secondary Outcome: Pregnancy Complications
Description: Reported complications during pregnancy, including spontaneous abortion, vaginal or uterine bleeding, emergency c-section and other complications
Time Frame: up to 60 weeks
Population: Women becoming pregnant during regular follow-up in the study (70 in Truvada group and 45 in placebo group)
Measure: Number; unit: participants
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 70 | 45
participants | 20 | 10

11. Secondary Outcome: Pill Counts and Participant Report of Adherence to Once-daily Pill Taking
Description: Pill counts and participant report of adherence to once-daily pill taking reported as mean days study product could have been used according to pill counts
Time Frame: Up to 52 weeks
Population: All randomized participants who completed at least one follow-up visit, excluding women found to have been infected at enrollment
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 1024 | 1032
percentage of days | 87 (0.20) | 89 (0.17)

12. Secondary Outcome: Participant Report of Change in Number of Sexual Partners
Description: Difference in mean number of reported sexual partners between final study visit and enrollment visit
Time Frame: Up to 52 weeks
Population: Women reporting on sexual behavior during follow-up
Measure: Mean (Standard Deviation); unit: mean number of sexual partners
Arm/Group | Truvada Arm | Placebo Arm
Number analyzed (Participants) | 977 | 989
mean number of sexual partners | -0.14 (0.60) [0 to 6] | -0.13 (0.79) [0 to 11]
Statistical Analysis 1: Comparison: Truvada Arm vs Placebo Arm; t-test for difference in change in number of sexual partners over time; Test type: Superiority or Other; p = 0.73, t-test, 2 sided; Mean Difference (Final Values) = .01

ADVERSE EVENTS:
Description: These data are from the safety population, which is a subset of the intent to treat (ITT) population, excluding those participants found to have been HIV infected at enrollment and participants who never received study product, returned all product unused, or never returned for a follow-up visit.
Arm/Group | Truvada Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 33/1025 | 23/1033
Other Adverse Events (participants affected / at risk) | 761/1025 | 749/1033
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Truvada Arm (N=1025) | Placebo Arm (N=1033)
anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
exomphalos (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
typhoid fever (Gastrointestinal disorders) | 2 (2) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
malaria (Infections and infestations) | 4 (4) | 3 (3)
pneumonia (Infections and infestations) | 1 (1) | 1 (1)
respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0)
influenza (Infections and infestations) | 1 (1) | 0 (0)
pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
wound (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
joint dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 2 (2) | 1 (1)
muscular weakness (Nervous system disorders) | 1 (1) | 0 (0)
neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
abortion (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
premature rupture of the membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
intentional overdose (Psychiatric disorders) | 1 (1) | 2 (2)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
removal of foreign body (Surgical and medical procedures) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Truvada Arm (N=1025) | Placebo Arm (N=1033)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 5 (6)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Exomphalos (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 5 (5)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 4 (4)
Abnormal vision (Eye disorders) | 1 (2) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 50 (52) | 32 (33)
Abdominal pain (Gastrointestinal disorders) | 27 (27) | 27 (27)
Vomiting (Gastrointestinal disorders) | 37 (38) | 12 (12)
Typhoid fever (Gastrointestinal disorders) | 24 (25) | 14 (17)
Gastroenteritis (Gastrointestinal disorders) | 21 (21) | 14 (16)
Diarrhoea (Gastrointestinal disorders) | 17 (18) | 17 (21)
Dyspepsia (Gastrointestinal disorders) | 11 (11) | 16 (17)
Toothache (Gastrointestinal disorders) | 13 (15) | 7 (7)
Gastritis (Gastrointestinal disorders) | 8 (8) | 11 (11)
Dysentery (Gastrointestinal disorders) | 7 (8) | 5 (5)
Flatulence (Gastrointestinal disorders) | 5 (5) | 6 (6)
Dental caries (Gastrointestinal disorders) | 2 (2) | 3 (3)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 17 (17) | 8 (8)
Malaise (General disorders) | 7 (8) | 11 (11)
Pain (General disorders) | 4 (4) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0)
Procedural pain (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Immune system disorders) | 30 (33) | 21 (21)
Pruritus allergic (Immune system disorders) | 11 (12) | 6 (6)
Conjunctivitis allergic (Immune system disorders) | 3 (3) | 9 (9)
Hypersensitivity (Immune system disorders) | 8 (8) | 2 (2)
Rhinitis allergic (Immune system disorders) | 1 (1) | 4 (5)
Allergic cough (Immune system disorders) | 2 (3) | 1 (1)
Allergic sinusitis (Immune system disorders) | 1 (1) | 0 (0)
Idiopathic urticaria (Immune system disorders) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 123 (154) | 121 (157)
Respiratory tract infection (Infections and infestations) | 96 (108) | 108 (125)
Vaginitis bacterial (Infections and infestations) | 67 (69) | 81 (81)
Candidiasis (Infections and infestations) | 60 (62) | 52 (57)
Chlamydial infection (Infections and infestations) | 35 (35) | 38 (39)
Urinary tract infection (Infections and infestations) | 23 (23) | 34 (38)
Nasopharyngitis (Infections and infestations) | 19 (21) | 36 (42)
Tonsillitis (Infections and infestations) | 23 (28) | 23 (26)
Tinea infection (Infections and infestations) | 18 (18) | 19 (22)
Pelvic inflammatory disease (Infections and infestations) | 16 (16) | 20 (20)
Vaginal infection (Infections and infestations) | 20 (23) | 12 (12)
Trichomoniasis (Infections and infestations) | 13 (13) | 16 (16)
Influenza (Infections and infestations) | 13 (14) | 14 (16)
Pneumonia (Infections and infestations) | 12 (13) | 13 (14)
Cervicitis (Infections and infestations) | 11 (11) | 10 (10)
Abscess (Infections and infestations) | 9 (9) | 8 (8)
Gonorrhoea (Infections and infestations) | 10 (10) | 5 (5)
Sinusitis (Infections and infestations) | 7 (7) | 2 (2)
Furuncle (Infections and infestations) | 5 (5) | 3 (4)
Tuberculosis (Infections and infestations) | 4 (4) | 2 (2)
Vulvovaginitis (Infections and infestations) | 4 (4) | 2 (2)
Wound infection (Infections and infestations) | 3 (3) | 3 (3)
Eye infection (Infections and infestations) | 3 (3) | 2 (2)
Oral herpes (Infections and infestations) | 4 (5) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Otitis externa (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 3 (3)
Helminthic infection (Infections and infestations) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Amoebiasis (Infections and infestations) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 1 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Extrapulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 5 (5) | 11 (11)
Joint sprain (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Human bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion of knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 199 (267) | 189 (257)
Aspartate aminotransferase increased (Investigations) | 134 (177) | 119 (147)
Alanine aminotransferase increased (Investigations) | 119 (162) | 110 (125)
Blood phosphorus increased (Investigations) | 93 (103) | 102 (121)
Blood creatinine increased (Investigations) | 70 (95) | 67 (79)
Liver function test abnormal (Investigations) | 26 (35) | 18 (19)
Blood bicarbonate decreased (Investigations) | 12 (13) | 20 (22)
Eosinophil count increased (Investigations) | 1 (1) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Glucose urine (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 1 (1)
Hormonal level abnormal (Investigations) | 1 (1) | 0 (0)
Renal function test abnormal (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (22) | 25 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (12)
Soft tissue injury (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 134 (153) | 148 (173)
Dizziness (Nervous system disorders) | 52 (56) | 45 (46)
Hypoaesthesia (Nervous system disorders) | 5 (6) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 4 (5) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 2 (3)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Muscular weakness (Nervous system disorders) | 1 (1) | 0 (0)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Vision blurred (Nervous system disorders) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 7 (7)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature rupture of the membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Somatoform disorder pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Intentional overdose (Psychiatric disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 19 (22) | 13 (14)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 17 (18) | 13 (13)
Metrorrhagia (Reproductive system and breast disorders) | 10 (10) | 14 (15)
Menorrhagia (Reproductive system and breast disorders) | 12 (12) | 9 (9)
Dysmenorrhoea (Reproductive system and breast disorders) | 8 (8) | 6 (6)
Genital ulceration (Reproductive system and breast disorders) | 10 (10) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 3 (3) | 4 (4)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 5 (5)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Premenstrual syndrome (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Coital bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Galacthorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital erosion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (10)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chloasma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Physical assault (Social circumstances) | 1 (1) | 0 (0)
Removal of foreign body (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Venous insufficiency (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes